CLINICAL TRIAL: NCT02828943
Title: Combined Inspiratory and Expiratory Muscle Training in Long-term Stroke
Brief Title: Ventilatory Muscle Training in Stroke
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Responsible Party: Principal Investigator, Elliot Roth, Medical Director of Patient Recovery Unit, Shirley Ryan AbilityLab
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STU00202271
Record Dates: First submitted 2016-07-06; First posted 2016-07-12 (Estimated); Last update posted 2019-01-17 (Actual); Status verified 2019-01

CONDITIONS: Stroke; Pulmonary Ventilation; Exercise Therapy
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- IMT with Low Resistance EMT (Active Comparator): The pressure loads can be adjusted at 2 cm H2O intervals for the Threshold IMT, up to 41 cm H2O, and 1 cm H2O intervals for the Threshold PEP, up to 20 cm H2O. For the comparator group, EMT will be set to 5 cm H2O, the lowest setting on the device. IMT training loads will be set to 30% of maximal inspiratory pressure for both groups. The patient will be blinded to the valve titration. Each training session will include one set of 10 repetitions with IMT followed by one set of 10 repetitions with low resistance EMT. Patients will be instructed to maintain a respiratory rate of 15-20 breaths/min without rest between repetitions. Participants will be monitored daily by phone and by self-reported log for completion of each training.
  Interventions: Behavioral: IMT with Low Resistance EMT
- IMT with High Resistance EMT (Experimental): The pressure loads can be adjusted at 2 cm H2O intervals for the Threshold IMT, up to 41 cm H2O, and 1 cm H2O intervals for the Threshold PEP, up to 20 cm H2O. EMT training loads in the experimental group will be set to 30% of maximal expiratory pressure. IMT training loads will be set to 30% of maximal inspiratory pressure for both groups. The patient will be blinded to the valve titration. Each training session will include one set of 10 repetitions with IMT followed by one set of 10 repetitions with high resistance EMT. Patients will be instructed to maintain a respiratory rate of 15-20 breaths/min without rest between repetitions. Participants will be monitored daily by phone and by self-reported log for completion of each training. At two weeks, participants will have a follow-up office visit to monitor progress and those that have completed 80% of their training sessions will increase their training to 40% of maximum inspiratory and expiratory pressures as tolerated.
  Interventions: Behavioral: IMT with High Resistance EMT

INTERVENTIONS:
Behavioral: IMT with High Resistance EMT
  Arms: IMT with High Resistance EMT
Behavioral: IMT with Low Resistance EMT
  Arms: IMT with Low Resistance EMT

SUMMARY:
The purpose of the present study is to determine the utility and effectiveness of combined inspiratory (IMT) and expiratory muscle training (EMT) in improving ventilatory function in people who are disabled by long-term stroke (greater than 8 months following onset) with hemiparesis or hemiplegia. xx subjects will be randomized into 2 parallel groups in which the experimental group will undergo combined IMT and high-resistance EMT and the comparison group will undergo IMT with low- resistance EMT. Both training techniques involve breathing through a tube with known amounts of resistance. Subjects will perform the breathing maneuvers for 10 repetitions, twice daily, 5 days per week for 4 weeks, in the home environment. Adherence will be monitored by reminder telephone calls at least weekly. Outcomes will be assessed using maximum inspiratory and expiratory pressures and standard pulmonary function testing.

DETAILED DESCRIPTION:
The purpose of the present study is to determine the utility and effectiveness of Expiratory Muscle Training in improving respiratory muscle strength in patients with chronic stroke, when combined with Inspiratory Muscle Training.

20 participants will be recruited from one site (Rehabilitation Institute of Chicago). All participants will give written informed consent before the enrollment in the study. Participants will be compensated for their participation.

Participants will participate in the study for one month. Maximum inspiratory and expiratory pressures will be measured in the seated position. Pulmonary function testing will also be performed in the seated position using a spirometer. Dyspnea will be assessed by the Medical Research Council (MRC) dyspnea scale.

The initial evaluation will consist of recording demographic information and conducting a comprehensive medical history, including: age, gender, race, marital status, education, employment, smoking history, ischemic stroke etiology, stroke severity with NIH Stroke Scale, and stroke location. This information may also be obtained from the RIC electronic medical record. Each subject will undergo a thorough neurologic assessment.

Study participants will be randomly assigned to one of two groups: the experimental group with high resistance EMT and the control group with low resistance EMT. The participants will be randomized to the two groups by an independent staff member at the time of enrollment based on the medical record number. Both groups will undergo IMT because IMT has been found to be effective improving MIP as well as FEV1 and FVC. The patients and those reading the pulmonary function tests will be blinded to the group assignment of each participant.

Upon enrollment in the study, respiratory muscle training will be completed twice daily for 5 days a week for 4 weeks. Training will be provided with the Threshold IMT (Respironics, Murrysville, PA) for inspiratory training and Threshold PEP (Respironics, Murrysville, PA) for expiratory training. The Threshold respiratory trainers are commercially available devices with a spring-loaded valve that provided resistance. The pressure loads can be adjusted at 2 cm H2O intervals for the Threshold IMT, up to 41 cm H2O, and 1 cm H2O intervals for the Threshold PEP, up to 20 cm H2O. EMT training loads in the experimental group will be set to 30% of maximal expiratory pressure while the control group EMT will be set to 5 cm H2O, the lowest setting on the device. IMT training loads will be set to 30% of maximal inspiratory pressure for both groups. The patient will be blinded to the valve titration. Each training session will include one set of 10 repetitions with IMT followed by one set of 10 repetitions with high resistance EMT or low resistance EMT. Patients will be instructed to maintain a respiratory rate of 15-20 breaths/min without rest between repetitions. Participants will be monitored daily by phone and by self-reported log for completion of each training. At two weeks, participants will have a follow-up office visit to monitor progress and those that have completed 80% of their training sessions will increase their training to 40% of maximum inspiratory and expiratory pressures as tolerated.

Each participant will undergo baseline measurement of maximal inspiratory and expiratory pressure and baseline pulmonary function tests as well as after 4 weeks of training. Three trials will be performed with the highest result of the three trials recorded.

ELIGIBILITY:
Inclusion Criteria:

1. History of Ischemic stroke
2. Stroke impairment 8 months or more
3. Hemiparesis in upper and/or lower limb
4. Ability to give informed consent
5. Ability to follow instructions for study procedures
6. Completed a standard multidisciplinary inpatient stroke rehabilitation program consisting of physical, occupational, and speech therapy sessions for at least 3 hours a day for 5 days a week for at least 2 weeks

Exclusion Criteria:

1. Neurological conditions other than stroke
2. Active concurrent exacerbation of cardiopulmonary disease
3. Presence of a tracheostomy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Maximum inspiratory pressure | 4 weeks
  Maximum inspiratory pressure

SECONDARY OUTCOMES:
Maximum expiratory pressure | 4 weeks
  Maximum expiratory pressure
Medical Research Council (MRC) dyspnea scale | 4 weeks
  Medical Research Council (MRC) dyspnea scale

CONTACTS AND LOCATIONS:
Locations (1):
- Shirley Ryan AbilityLab, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided